CLINICAL TRIAL: NCT05249387
Title: Characterization of Bovine Adrenal Medulla (BAM8-22) as a New Surrogate Model of Non-histaminergic Itch
Brief Title: Characterization of Bovine Adrenal Medulla as a New Surrogate Model of Non-histaminergic Itch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Giulia Erica Aliotta, Principal Investigator, PhD fellow, Aalborg University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20190062 5th project
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Itch
MeSH Terms: conditions — Pruritus | interventions — A 967079

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-967079 Injections + BAM8-22 (Experimental)
  Interventions: Drug: A-967079 and BAM8-22 application; Drug: A-967079 and BAM8-22 application after 5 minutes.
- A-967079 Injections and vehicle (Experimental)
  Interventions: Drug: A-967079 application.; Drug: Vehicle and BAM8-22 application.

INTERVENTIONS:
Drug: A-967079 and BAM8-22 application — A-967079 solution (in PBS 0.5 mg/ml, subcutaneous injection of 0.1ml) and BAM8-22 with inactivate cowhage spicules 20 µl of BAM8-22 will be applied to a previously determined area on the volar forearm using inactivate cowhage spicules
  Arms: A-967079 Injections + BAM8-22
Drug: A-967079 and BAM8-22 application after 5 minutes. — A-967079 solution (in PBS 0.5 mg/ml, subcutaneous injection of 0.1ml). BAM8-22 with inactivate cowhage spicules 20 µl of BAM8-22 will be applied 5 minutes after to a previously determined area on the volar forearm using inactivate cowhage spicules
  Arms: A-967079 Injections + BAM8-22
Drug: A-967079 application. — A-967079 solution (in PBS 0.5 mg/ml, subcutaneous injection of 0.1ml) will be applied to a previously determined area on the volar forearm
  Arms: A-967079 Injections and vehicle
Drug: Vehicle and BAM8-22 application. — Vehicle (in PBS, subcutaneous injection of 0.1ml) and BAM8-22 with inactivate cowhage spicules 20 µl of BAM8-22 will be applied to a previously determined area on the volar forearm using inactivate cowhage spicules
  Arms: A-967079 Injections and vehicle

SUMMARY:
With this experiment, the experimenter wish evaluate the role of TRPA1 on non-histaminergic itch induced by BAM8-22

DETAILED DESCRIPTION:
With this experiment, the experimenter wish evaluate the role of TRPA1 on non-histaminergic itch induced by BAM8-22 2 (Bovine Adrenal Medulla), which is found naturally in the human body and which has proved to evoke itch. To evaluate the role of TRPA1 it will be used a TRPA1 antagonist (A-967079)

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids or other drugs
* Previous or current history of neurological, dermatological, immunological musculoskeletal, cardiac disorder or mental illnesses that may affect the results (e.g. neuropathy, muscular pain in the upper extremities, etc.)
* Moles, wounds, scars or tattoos in the area to be treated or tested
* Lack of ability to cooperate •
* Current use of medications that may affect the trial such as antihistamines and pain killers.
* Skin diseases
* Consumption of alcohol or painkillers 24 hours before the study days and between these - Acute or chronic pain •
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
superficial blood perfusion | change from baseline, up to 10 minutes after the application
  is measured by a speckle contrast imager (FLPI, Moor Instruments, England)
Warm Detection Threshold, and Heat Pain threshold | change from baseline, up to 10 minutes after the application
  he tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Cold Detection Threshold and Cold Pain threshold | change from baseline, up to 10 minutes after the application
  the tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Pain supra-threshold heat Stimuli | change from baseline, up to 10 minutes after the application
  the tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Alloknesis | change from baseline, up to 10 minutes after the application
  s measured by using a mildy pruritic, non-painful von Frey filaments of a predetermined intensity (generally 5-30 milliNewton of force)
mechanical pain threshold and sensitivity | change from baseline, up to 10 minutes after the application
  is performed using a pin-prick set (Aalborg University). The set consists of 8 needles each having a diameter of 0,6 mm and different force applications
itch rating | change from baseline, up to 10 minutes after the application
  the subject will rate the itch for 10 minutes by using a visual analog scale (VAS) on a tablet. this scale goes from 0 to 100. 0 indicates "no itch" and 100 indicates "worst imaginable itch"

SECONDARY OUTCOMES:
pain rating | change from baseline, up to 10 minutes after the application
  the subject will rate the pain for 10 minutes by using a visual analog scale (VAS) on a tablet. this scale goes from 0 to 100. 0 indicates "no pain" and 100 indicates "worst imaginable pain"

CONTACTS AND LOCATIONS:
Locations (1):
- Giulia Erica Aliotta, Aalborg, Denmark